CLINICAL TRIAL: NCT01071837
Title: A Phase II, Randomized, Open-label, Multi-centre Study of Weekly APG101 + Reirradiation Versus Reirradiation in the Treatment of Patients With First or Second Progression of Glioblastoma
Brief Title: APG101 in Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apogenix GmbH (Industry)
Responsible Party: Sponsor
Organization: Apogenix AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG101_CD_002
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — APG101; Recombinant Fusion Proteins; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Re-Irradiation (Active Comparator): 33% of the patients will be randomized to reirradiation (RT) alone. They will receive 36 Gy (2 Gy per fraction)
  Interventions: Procedure: Blood drawing
- Re-Irradiation + APG101 (Experimental): 66% of the patients will be randomized to reirradiation (RT) + 400 mg APG101 weekly. They will receive 36 Gy (2 Gy per fraction) and 400 mg APG101 weekly as an intravenous infusion
  Interventions: Drug: APG101

INTERVENTIONS:
Drug: APG101 — 400mg weekly as intravenous infusion
  Other Names: Recombinant fusion protein
  Arms: Re-Irradiation + APG101
Procedure: Blood drawing — Blood drawings, e.g. for safety labs, abdominal ultrasound, ECG. Re-Irradiation is not considered a study procedure, but standard of care (inclusion criterion)
  Arms: Re-Irradiation

SUMMARY:
This is a phase II study of APG101 + reirradiation (RT) versus reirradiation. Patients suffering from a malignant brain tumor called glioblastoma having a first or second progression can be included. They will be randomized to RT or RT + APG101.

APG101 is a fusion protein (similar to an antibody) and will be administered as a weekly infusion. Patients can stay in this study as long as they benefit from the participation (no fixed end).

In this trial, 30-35 sites in Germany, Austria and Russia take part.

DETAILED DESCRIPTION:
In this phase II trial, patients with a recurrence / progression of glioblastoma (first or second progression) either not being eligible for tumour resection or having macroscopic residual tumour after resection of the recurrence can be included (tumor size must 1-4 cm in T1-weighted MRI). They must be candidates for a re-irradiation and will then be randomized in a 1:2 ratio to re-irradiation alone or re-irradiation + 400mg APG101 as a weekly intravenous infusion.

Radiotherapy (RT) is considered standard of care and not a study procedure. As prior therapies, a first radiotherapy (maximal dose of 60 Gy; at least 8 months since the end of preirradiation), a prior surgery (at least for histology) and at least one Temozolomide-containing chemotherapy are mandatory; patients with prior treatment with bevacizumab, iodine seeds and/or brachytherapy are not eligible. The patients' steroid dose must be stable or decreasing upon inclusion.

The number of patients to be included in this study is up to 83 (depending on the statistical 2-step SIMON design).

Primary objective: 6 months rate of progression free survival (PFS6). Subjects can participate in this study as long as a clinical benefit is considered by the treating physician.

MRI tumour imaging will be carried out every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a recurrence / progression of glioblastoma either not being eligible for tumour resection or having macroscopic residual tumour after resection of the recurrence
* Diagnosis of glioblastoma must be proven histologically and progress must be documented by MRI. MRI images must not be older than 2 weeks before first dosing/start of RT
* Not more than two prior therapy regimens including one or two resections, one or two chemotherapies of which one must have been TMZ-containing and one radiotherapy (RT) for the brain tumour
* Previous irradiation therapy of the primary tumour with a maximal dose of 60 Gy; at least 8 months since the end of preirradiation
* Candidate for reirradiation with recurrent tumour visible on MRI-T1 (Gd) and with the largest diameter measuring 1 cm to 4 cm
* Informed consent
* Age at least 18 years, smoking or non-smoking, of any ethnic origin
* Karnofsky performance index (KPI) ≥ 60%
* Neutrophile counts > 1500/μl / Platelet counts > 80.000/μl / Haemoglobin > 10 g/dl / Serum creatinine < 1.5-fold upper normal range / Bilirubin, AST or ALT < 2,5-fold upper normal range unless attributed to anticonvulsants / Alkaline phosphatase < 2,5-fold upper normal range
* Adequate contraception
* Stable or decreasing treatment with steroids within 5 days before treatment start

Exclusion Criteria:

* More than one RT of brain, prior first radiotherapy with more than 60 Gy
* Cumulative total dose on the optical chiasm >54 Gy for 2 Gy/fraction, α/β=2
* Prior treatment with bevacizumab, iodine seeds and/or brachytherapy
* Unable to undergo MRI
* Past medical history of diseases with poor prognosis according to the judgement of the Investigator, e.g. severe coronary heart disease, severe diabetes, immune deficiency, residual deficits after stroke, severe mental retardation
* HIV or hepatitis infection
* Pregnancy or breast feeding
* Treatment within any other clinical trial parallel to the treatment phase of the current study or within 30 days before inclusion
* Known active coronary artery disease, significant cardiac arrhythmias or severe congestive heart failure (NYHA class III - IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
6 months rate of progression free survival (PFS6) | 6 month

SECONDARY OUTCOMES:
Safety and tolerability of APG101 | ongoing during study
Progression-free survival | until progression of underlying disease
Objective response rates (OR) | ongoing during study
Duration of response (DR) in responders | ongoing during study
Overall survival | until study and after end of study (by 8-weekly phone calls)
Quality of life | ongoing during study
Cognitive function | ongoing during study

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, MD, Study Director — University Hospital Heidelberg, Dept. of Neurooncology, Germany
Locations (21):
- Austria (4):
  - Medizinische Universität Graz, Universitätsklinik für Neurologie Landeskrankenhaus Graz, Graz
  - Universitätsklinik für Neurologie, Landeskrankenhaus Innsbruck, Innsbruck
  - Landesnervenklinik Wagner-Jauregg, Innere Medizin mit Neuroonkologie, Linz
  - Allgemeines Krankenhaus der Stadt Wien, Klinische Onkologie, Vienna
- Germany (17):
  - Charite Universitätsmedizin Berlin, Klinik für Neurochirugie, Berlin
  - Neurologische Universitätsklinik am Knappschaftskrankenhaus, Bochum
  - Neurologische Universitätsklinik Bonn, Schwerpunkt klinische Neuroonkologie, Bonn
  - Universitätsklinik Dresden, Klinik und Poliklinik für Neurochirurgie, Dresden
  - Klinikum Frankfurt/Oder, Klinik für Strahlentherapie/Radioonkologie, Frankfurt (Oder)
  - Universitätsklinik Hamburg, Klinik für Neurochirugie, Hamburg
  - Universitätsklinik Heidelberg, Abteilung Neuroonkologie, Heidelberg
  - Universität Leipzig, Klinik für Strahlentherapie, Leipzig
  - Universitätsmedizin Mannheim, Klinik für Neurochirurgie, Mannheim
  - Philipps-Universität Marburg, Klinik für Neurologie, Marburg
  - LMU München, Klinik und Poliklinik für Strahlentherapie und Radioonkologie, Campus Großhadern & Campus Innenstadt, München
  - Klinik und Poliklinik für Strahlentherapie/Radiologische Onkologie, Klinikum rechts der Isar, TU München, München
  - Städt. Kliniken München GmbH, Klinikum Bogenhausen, Abt. Neurochirurgie, München
  - Klinik und Poliklinik der Universität Regensburg, Im Bezirksklinikum, Regensburg
  - Klinikum Stuttgart, Neurozentrum Neurochirurgie, Stuttgart
  - Universitätsklinikum Tuebingen, Strahlenonkologie, Tübingen
  - Uniklinik Ulm, Klinik für Strahlentherapie und Radioonkologie, Ulm